CLINICAL TRIAL: NCT02840617
Title: A Pilot and Feasibility Study of Indocyanine Green-based Fluorescence Imaging in Localization of Prostate Cancer and Metastatic Lymph Nodes
Brief Title: ICG-based Fluorescence Imaging in Localization of Prostate Cancer and Metastatic Lymph Nodes
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Rongqin Zheng, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: sysu160511
Record Dates: First submitted 2016-07-05; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: ICG; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Indocyanine Green

ARMS (1):
- ICG injection group (Experimental): ICG will be intravenously administered over a 10 second period immediately after the patient was anesthetized. The fluorescence will be performed during and after the surgery, respectively.
  Interventions: Drug: Indocyanine Green (ICG)

INTERVENTIONS:
Drug: Indocyanine Green (ICG)
  Other Names: ICG

SUMMARY:
This study aims to evaluate the feasibility of indocyanine green (ICG)-based fluorescence imaging in the detection of prostate tumors and metastatic lymph nodes. By correlating the ICG fluorescence patterns with pathologically confirmed tumor and nodal status, it would be possible to use fluorescence navigation system in helping prostate biopsy and lymph node dissection in the future.

DETAILED DESCRIPTION:
The investigators will conduct an in vivo and in vitro pilot study in order to evaluate the diagnostic performance of fluorescence in the detection of prostate cancer and metastatic lymph nodes. All the patients included in this study will receive a radical prostatectomy after intravenous injection of 0.4 mg/Kg of ICG. ICG will be administered immediately after the patient is anesthetized. The fluorescence analysis will be performed intraoperatively by laparoscopic imaging and after surgery by hand-held imaging. The prostate or lymph nodes specimen with or without fluorescence signal will be sent to the Department of Pathology for pathological analysis. The histopathological procedure will be performed without knowledge of fluorescence analysis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer;
* Able to accept total prostatectomy;
* Patient has given its informed consent.

Exclusion Criteria:

* Allergic to ICG or iodine;
* High-grade hepatic insufficiency
* refuse attending the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity of the ICG-based fluorescence to detect prostate cancer | 1 week post-surgery
  sensitivity (true positive) and specificity (true negative) of the ICG-based fluorescence to detect prostate cancer in vivo and in vitro compared to histological analysis

SECONDARY OUTCOMES:
sensitivity and specificity of the ICG-based fluorescence imaging to detect metastatic lymph nodes | 1 week post-surgery
  sensitivity (true positive) and specificity (true negative) of the ICG-based fluorescence to detect metastatic lymph nodes in vivo and in vitro compared to histological analysis

CONTACTS AND LOCATIONS:
Overall Officials: Rongqin Zheng RQ Zheng, doctor, Study Chair — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The department of Ultrasound, the third affiliated hospital of Sun Yat-son University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Greco F, Cadeddu JA, Gill IS, Kaouk JH, Remzi M, Thompson RH, van Leeuwen FW, van der Poel HG, Fornara P, Rassweiler J. Current perspectives in the use of molecular imaging to target surgical treatments for genitourinary cancers. Eur Urol. 2014 May;65(5):947-64. doi: 10.1016/j.eururo.2013.07.033. Epub 2013 Aug 7. PMID 23957947